CLINICAL TRIAL: NCT01133522
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 145 in Subjects With Hyperlipidemia on Stable Doses of a Statin
Brief Title: Ascending Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Evolocumab (AMG 145) in Adults With Hyperlipidemia on Stable Doses of a Statin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20080398
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Results first posted 2015-10-22 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Hyperlipidemia
Keywords: AMG145; Multiple Dose; Statin; Ascending
MeSH Terms: conditions — Hyperlipidemias | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evolocumab (Experimental): Participants received one of 5 dose levels of evolocumab administered as multiple subcutaneous doses.
  Interventions: Biological: Evolocumab
- Placebo (Placebo Comparator): Participants received matching placebo dose regimens by subcutaneous injection.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: Evolocumab
Biological: Placebo — Administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of multiple doses of evolocumab when given as an add-on to stable statin therapy.

DETAILED DESCRIPTION:
Participants receiving low-to-moderate-dose statins were randomized in a 1:3 ratio to receive subcutaneous placebo or evolocumab and enrolled sequentially into one of 5 dose-escalation cohorts:

1. Evolocumab 14 mg/placebo once weekly (QW) × 6 doses
2. Evolocumab 35 mg/placebo once weekly (QW) × 6 doses
3. Evolocumab 140 mg/placebo every 2 weeks (Q2W) × 3 doses
4. Evolocumab 280 mg/placebo every 2 weeks (Q2W) × 3 doses
5. Evolocumab 420 mg/placebo every 4 weeks (Q2W) × 2 doses.

Participants receiving high-dose statins were randomized 1:3 to receive subcutaneous placebo or evolocumab 140 mg every 2 weeks × 3 doses (Cohort 6).

Participants diagnosed with familial hypercholesterolemia (HeFH) were randomized 1:2 to receive subcutaneous placebo or evolocumab 140 mg every 2 weeks × 3 doses (Cohort 7).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 to 70 years (inclusive) at the time of screening with hyperlipidemia
* Body mass index (BMI) ≥18 and ≤ 35 kg/m^2 at the time of screening
* Low-density lipoprotein cholesterol (LDL-C) level of 70-220 mg/dL (inclusive) at screening as measured by direct assay
* For Cohorts 1-5: On a stable dose of rosuvastatin (Crestor) < 40 mg/day, atorvastatin (Lipitor) < 80 mg/day, or simvastatin (Zocor) 20-80 mg/day for ≥ 1 month prior to enrollment and expected to remain on this dose for the remainder of the study
* For Cohort 6: On a stable dose of rosuvastatin (Crestor) 40 mg/day or atorvastatin (Lipitor) 80 mg/day for ≥ 1 month prior to enrollment and expected to remain on this dose for the remainder of the study
* For Cohort 7: Diagnosis of heterozygous familial hypercholesterolemia, based on a score of ≥ 9 points using the World health Organization (WHO) criteria

Exclusion Criteria:

* Diagnosis of homozygous familial hypercholesterolemia
* History of heart failure, coronary artery bypass graft, or cardiac arrhythmia
* History of acute coronary syndrome (e.g. myocardial infarction, hospitalization for unstable angina) or percutaneous coronary intervention, within 12 months prior to enrollment
* Planned cardiac surgery or revascularization
* Known aortic, peripheral vascular or cerebrovascular disease (including history of stroke or transient ischemic attack)
* Diabetes mellitus with any of the following:

  1. known microvascular or macrovascular disease
  2. HbA1c > 8.0% at screening
  3. use of any hypoglycemic medication other than metformin
* Uncontrolled hypertension (systolic blood pressure ≥ 150 or diastolic blood pressure ≥ 90 mmHg) either on or off therapy at screening or at baseline

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2011-09-14 (Actual); Study Completion 2011-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Dias CS, Shaywitz AJ, Wasserman SM, Smith BP, Gao B, Stolman DS, Crispino CP, Smirnakis KV, Emery MG, Colbert A, Gibbs JP, Retter MW, Cooke BP, Uy ST, Matson M, Stein EA. Effects of AMG 145 on low-density lipoprotein cholesterol levels: results from 2 randomized, double-blind, placebo-controlled, ascending-dose phase 1 studies in healthy volunteers and hypercholesterolemic subjects on statins. J Am Coll Cardiol. 2012 Nov 6;60(19):1888-98. doi: 10.1016/j.jacc.2012.08.986. Epub 2012 Oct 17. PMID 23083772
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled hypercholesterolemic adults receiving stable statin therapy (7 cohorts: 5 on low-to-moderate-dose statins, 1 on high-dose statin therapy, and 1 with heterozygous familial hypercholesterolemia (HeFH) (score ≥9, World Health Organization criteria). First patient enrolled 28 June 2010. Last patient enrolled 24 June 2011.
Pre-assignment Details: Participants receiving low-to-moderate-dose statins were randomized 1:3 to placebo or evolocumab and sequentially assigned to 1 of 5 dose-escalation cohorts. The high-dose statin and HeFH cohorts were randomized 1:3 and 1:2 respectively to placebo or evolocumab. Placebo participants were pooled for the 5 dose-escalation cohorts.
Groups:
- Placebo: Cohorts 1-5 Combined: Participants on low-to-moderate dose statin therapy received placebo subcutaneous injections matching active investigational product in volume and frequency.
- Evolocumab 14 mg QW × 6: Cohort 1: Participants on low-to-moderate-dose stain therapy received evolocumab 14 mg subcutaneous injection once weekly (QW) for 6 weeks.
- Evolocumab 35 mg QW × 6: Cohort 2: Participants on low-to-moderate-dose statin therapy received evolocumab 35 mg subcutaneous injection once weekly for 6 weeks.
- Evolocumab 140 mg Q2W × 3: Cohort 3: Participants on low-to-moderate-dose statin therapy received evolocumab 140 mg subcutaneous injection every 2 weeks (Q2W) for 6 weeks.
- Evolocumab 280 mg Q2W × 3: Cohort 4: Participants on low-to-moderate-dose statin therapy received evolocumab 280 mg subcutaneous injection every 2 weeks for 6 weeks.
- Evolocumab 420 mg Q4W × 2: Cohort 5: participants on low-to-moderate-dose statin therapy received evolocumab 420 mg subcutaneous injection every 4 weeks (Q4W) for 8 weeks.
- High Dose Statin - Placebo: Cohort 6: Participants on high-dose statin therapy received placebo subcutaneous injection every 2 weeks for 6 weeks.
- High Dose Statin - Evolocumab 140 mg Q2W × 3: Cohort 6: Participants on high-dose statin therapy received evolocumab 140 mg subcutaneous injection every 2 weeks for 6 weeks.
- HeFH - Placebo: Cohort 7: Participants diagnosed with HeFH received placebo subcutaneous injection every 2 weeks for 6 weeks.
- HeFH - Evolocumab 140 mg Q2W × 3: Cohort 7: Participants diagnosed with HeFH received evolocumab 140 mg subcutaneous injection every 2 weeks for 6 weeks.
Period: Overall Study
Arm/Group | Placebo | Evolocumab 14 mg QW × 6 | Evolocumab 35 mg QW × 6 | Evolocumab 140 mg Q2W × 3 | Evolocumab 280 mg Q2W × 3 | Evolocumab 420 mg Q4W × 2 | High Dose Statin - Placebo | High Dose Statin - Evolocumab 140 mg Q2W × 3 | HeFH - Placebo | HeFH - Evolocumab 140 mg Q2W × 3
Started | 10 | 7 | 6 | 7 | 7 | 6 | 2 | 9 | 2 | 4
Received Treatment | 10 | 6 | 6 | 6 | 6 | 6 | 2 | 9 | 2 | 4
Completed | 10 | 6 | 6 | 6 | 6 | 6 | 2 | 9 | 2 | 4
Not Completed | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (all participants who received at least 1 dose of study drug).
Groups:
- Evolocumab 14 mg QW × 6: Cohort 1: Participants on low-to-moderate-dose stain therapy received evolocumab 14 mg subcutaneous injection once weekly for 6 weeks.
- Evolocumab 140 mg Q2W × 3: Cohort 3: Participants on low-to-moderate-dose statin therapy received evolocumab 140 mg subcutaneous injection every 2 weeks for 6 weeks.
- Evolocumab 420 mg Q4W × 2: Cohort 5: participants on low-to-moderate-dose statin therapy received evolocumab 420 mg subcutaneous injection every 4 weeks for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Evolocumab 14 mg QW × 6 | Evolocumab 35 mg QW × 6 | Evolocumab 140 mg Q2W × 3 | Evolocumab 280 mg Q2W × 3 | Evolocumab 420 mg Q4W × 2 | High Dose Statin - Placebo | High Dose Statin - Evolocumab 140 mg Q2W × 3 | HeFH - Placebo | HeFH - Evolocumab 140 mg Q2W × 3 | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 2 | 9 | 2 | 4 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (7.5) | 61.3 (4.0) | 63.7 (6.3) | 56.2 (7.3) | 56.3 (8.6) | 53.8 (4.9) | 62.0 (1.4) | 58.2 (7.6) | 54.5 (10.6) | 45.0 (15.1) | 56.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 1 | 3 | 4 | 3 | 1 | 3 | 1 | 0 | 26
  Male | 4 | 2 | 5 | 3 | 2 | 3 | 1 | 6 | 1 | 4 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 9 | 6 | 6 | 4 | 6 | 3 | 2 | 7 | 2 | 2 | 47
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 7
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Japanese | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aborigine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Low-Density Lipoprotein Cholesterol (LDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 108.9 (21.9) | 126.7 (22.1) | 106.5 (29.4) | 113.7 (14.5) | 105.8 (17.0) | 120.3 (33.0) | 99.0 (31.1) | 100.2 (25.5) | 168.5 (57.3) | 134.5 (31.1) | 114.1 (27.8)
Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) Concentration [Mean (Standard Deviation); unit: ng/mL] | 429.0 (93.1) | 491.2 (157.9) | 399.8 (116.7) | 384.8 (88.0) | 373.7 (96.0) | 459.0 (163.4) | 382.5 (82.7) | 486.6 (214.0) | 478.5 (94.0) | 396.0 (86.4) | 432.0 (133.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The relationship of each adverse event to the investigational product was assessed by the investigator.
  A serious adverse event (SAE) is defined as an adverse event that
  * is fatal
  * is life threatening (places the subject at immediate risk of death)
  * requires in-patient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * is a congenital anomaly/birth defect
  * other significant medical hazard.
Time Frame: From the first dose of study drug until Day 85
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Evolocumab 14 mg QW × 6 | Evolocumab 35 mg QW × 6 | Evolocumab 140 mg Q2W × 3 | Evolocumab 280 mg Q2W × 3 | Evolocumab 420 mg Q4W × 2 | High Dose Statin - Placebo | High Dose Statin - Evolocumab 140 mg Q2W × 3 | HeFH - Placebo | HeFH - Evolocumab 140 mg Q2W × 3
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 2 | 9 | 2 | 4
participants
  Any adverse event | 7 | 2 | 5 | 4 | 6 | 3 | 1 | 7 | 1 | 1
  Treatment-related adverse events | 1 | 1 | 0 | 1 | 6 | 0 | 1 | 2 | 0 | 0
  Serious adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Discontinuations due to adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Deaths on study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Evolocumab
Description: Serum concentrations of evolocumab were measured by a validated enzyme-linked immunosorbent assay (ELISA). The lower limit of quantification (LLOQ) was 800 ng/mL.
Time Frame: Day 1, predose and Days 4, 8, 15, 22, 29, 36, 40, 43, 50, 57, 64, 71, 78, and 85
Population: The Pharmacokinetic analysis set consisted of all participants for whom at least 1 pharmacokinetic parameter or endpoint could be adequately estimated. Serum evolocumab concentrations were not detectable in Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Evolocumab 14 mg QW × 6 | Evolocumab 35 mg QW × 6 | Evolocumab 140 mg Q2W × 3 | Evolocumab 280 mg Q2W × 3 | Evolocumab 420 mg Q4W × 2 | High Dose Statin - Evolocumab 140 mg Q2W × 3 | HeFH - Evolocumab 140 mg Q2W × 3
Number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 9 | 4
μg/mL |  |  | 20.3 (13.2) | 62.8 (22.7) | 63.6 (11.2) | 16.3 (10.8) | 14.7 (2.9)

3. Primary Outcome: Number of Participants With Anti-Evolocumab Antibodies
Description: Serum samples were analyzed by an electrochemiluminescence (ECL)-based immunoassay for anti-evolocumab binding antibodies. Positive samples were subsequently tested in a receptor-ligand binding bioassay for anti-evolocumab neutralizing antibodies
Time Frame: From the first dose of study drug until Day 85
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Evolocumab 14 mg QW × 6 | Evolocumab 35 mg QW × 6 | Evolocumab 140 mg Q2W × 3 | Evolocumab 280 mg Q2W × 3 | Evolocumab 420 mg Q4W × 2 | High Dose Statin - Placebo | High Dose Statin - Evolocumab 140 mg Q2W × 3 | HeFH - Placebo | HeFH - Evolocumab 140 mg Q2W × 3
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 2 | 9 | 2 | 4
participants
  Binding Antibodies | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Neutralizing Antibodies | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Evolocumab
Description: Area under the unbound evolocumab serum concentration-time curve from time of last dose to time of last quantifiable concentration following the last dose of evolocumab.
Time Frame: Day 29 predose (last dose for Cohorts 3-7) and Days 36 (predose for Cohorts 1 and 2), 40, 43, 50, 57, 64, 71, 78, and 85
Population: Pharmacokinetic analysis set with available data
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Evolocumab 14 mg QW × 6 | Evolocumab 35 mg QW × 6 | Evolocumab 140 mg Q2W × 3 | Evolocumab 280 mg Q2W × 3 | Evolocumab 420 mg Q4W × 2 | High Dose Statin - Evolocumab 140 mg Q2W × 3 | HeFH - Evolocumab 140 mg Q2W × 3
Number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 8 | 4
day*μg/mL |  |  | 226 (249) | 1200 (634) | 903 (280) | 181 (157) | 165 (69)

5. Secondary Outcome: Percent Change From Baseline to End of the Dosing Interval in LDL-C
Time Frame: Baseline and Day 43 for QW and Q2W groups or Day 57 for Q4W group
Population: Participants with non-missing data
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Evolocumab 14 mg QW × 6 | Evolocumab 35 mg QW × 6 | Evolocumab 140 mg Q2W × 3 | Evolocumab 280 mg Q2W × 3 | Evolocumab 420 mg Q4W × 2 | High Dose Statin - Placebo | High Dose Statin - Evolocumab 140 mg Q2W × 3 | HeFH - Placebo | HeFH - Evolocumab 140 mg Q2W × 3
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 2 | 9 | 2 | 4
percent change | 3.14 (33.73) | -23.79 (21.57) | -51.76 (18.29) | -69.58 (18.13) | -74.65 (3.47) | -62.01 (11.43) | -3.01 (3.09) | -61.82 (17.67) | -4.89 (0.82) | -62.91 (16.04)

6. Secondary Outcome: Percent Change From Baseline to End of the Dosing Interval in PCSK9
Description: Serum PCSK9 concentrations were determined by using a qualified enzyme-linked immunosorbent assay (ELISA). The lower limit of quantification (LLOQ) was 15 ng/mL.
Time Frame: Baseline and Day 43 for QW and Q2W groups or Day 57 for Q4W group
Population: Participants with non-missing data
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Evolocumab 14 mg QW × 6 | Evolocumab 35 mg QW × 6 | Evolocumab 140 mg Q2W × 3 | Evolocumab 280 mg Q2W × 3 | Evolocumab 420 mg Q4W × 2 | High Dose Statin - Placebo | High Dose Statin - Evolocumab 140 mg Q2W × 3 | HeFH - Placebo | HeFH - Evolocumab 140 mg Q2W × 3
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 2 | 9 | 2 | 4
percent change | 6.00 (25.49) | -42.07 (16.99) | -64.46 (3.70) | -70.42 (16.05) | -91.49 (6.45) | -32.72 (29.41) | 43.60 (51.39) | -62.50 (18.33) | 36.76 (12.54) | -68.52 (10.67)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until Day 85
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Evolocumab 14 mg QW × 6 | Evolocumab 35 mg QW × 6 | Evolocumab 140 mg Q2W × 3 | Evolocumab 280 mg Q2W × 3 | Evolocumab 420 mg Q4W × 2 | High Dose Statin - Placebo | High Dose Statin - Evolocumab 140 mg Q2W × 3 | HeFH - Placebo | HeFH - Evolocumab 140 mg Q2W × 3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/9 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 7/10 | 2/6 | 5/6 | 4/6 | 6/6 | 3/6 | 1/2 | 7/9 | 1/2 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Evolocumab 14 mg QW × 6 (N=6) | Evolocumab 35 mg QW × 6 (N=6) | Evolocumab 140 mg Q2W × 3 (N=6) | Evolocumab 280 mg Q2W × 3 (N=6) | Evolocumab 420 mg Q4W × 2 (N=6) | High Dose Statin - Placebo (N=2) | High Dose Statin - Evolocumab 140 mg Q2W × 3 (N=9) | HeFH - Placebo (N=2) | HeFH - Evolocumab 140 mg Q2W × 3 (N=4)
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipoma excision (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.